CLINICAL TRIAL: NCT03069625
Title: Sit-to-stand Test Use in Children and Adolescents With Cystic Fibrosis : Correlations With 6-Minute Walking Test, Quadriceps and Respiratory Muscle Strength and Health Related Quality of Life
Brief Title: Sit-to-stand Test in Cystic Fibrosis Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier du Havre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 2016-A01377-44
Record Dates: First submitted 2017-02-16; First posted 2017-03-03 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-05

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Exercise Testing; Muscular strength; Pediatrics; Quality of life
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sit-to-stand test (Experimental): Children and adolescents will perform 2 STS tests. First one is used to eliminate learning effect. Number of repetitions will be noted at the end of the second test.
  Interventions: Behavioral: Sit-to-stand test
- 6-Minute Walk Test (Active Comparator): Children and adolescents will perform 2 6MWT tests. First one is used to eliminate learning effect. Number of repetitions will be noted at the end of the second test.
  Interventions: Behavioral: 6-Minute Walk Test

INTERVENTIONS:
Behavioral: Sit-to-stand test — CF young patients will perform 2 STS tests. Number of repetitions, cardio-respiratory response and physiological adaptations during the second test will be monitored.
  Arms: Sit-to-stand test
Behavioral: 6-Minute Walk Test — CF young patients will perform 2 6MWT tests. Number of repetitions, cardio-respiratory response and physiological adaptations during the second test will be monitored.
  Arms: 6-Minute Walk Test

SUMMARY:
Cystic fibrosis (CF) is a chronic hereditary respiratory disease. Exercise testing is part of CF patients regular assessment.

Cardio-Pulmonary Exercise Testing (CPET) is currently considered as the gold standard to assess physical capacities. However, simple field tests are emerging. These tests are easier to perform especially in a population of CF children and adolescents.

The 1minute Sit-To-Stand test have recently been evaluated in CF adults. This test correlates with maximal oxygen consumption during CPET.

The investigators hypothesized that this test also correlates with 6-Minute Walking distance (during a 6-min Walk Test), quadriceps strength, respiratory muscles strength and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Cystic Fibrosis
* Exacerbation-free last month before inclusion

Exclusion Criteria:

* Cardiovascular, neurological or musculoskeletal contra-indications to exercise testing
* Other respiratory disease (kyphoscoliosis, asthma ...)
* Exacerbation
* Unability to carry out field tests

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-24 (Actual)

PRIMARY OUTCOMES:
Correlation between number of repetitions (STS Test) and 6-Minute Walking Distance | This outcome will be measured after both tests realization up to 15 minutes.
  Comparison between the results of these two submaximal exercise tests

SECONDARY OUTCOMES:
Correlation between number of repetitions (STS test) and Maximal Inspiratory Pressure (MIP) | MIP will be measured after inclusion in the hour before field tests realization.
  MIP will be assessed using a microRPM Puma manometer.
Correlation between number of repetitions (STS test) and Maximal Expiratory Pressure (MEP) | MEP will be measured after inclusion in the hour before field tests realization.
  MEP will be assessed using a MicroRPM Puma manometer.
Correlation between number of repetitions (STS Test) and health-related quality of life | HRQoL testing will be carried out after inclusion in the hour before field tests realization.
  HRQoL will be measured by the Cystic Fibrosis Questionnaire
Correlation between number of repetitions (STS Test) and quadriceps strength. | Quadriceps strength will be assessed after inclusion in the hour before field tests realization.
  Quadriceps strength will be assessed by handheld dynamometry using a MicroFet II dynamometer.
Correlation between number of repetitions (STS Test) and forced vital capacity (FVC) | Spirometric test will be carried out before field tests realization.
  FVC will be assessed with non invasive spirometry.
Correlation between number of repetitions (STS Test) and forced expiratory volume in 1 second (FEV1) | Spirometric test will be carried out in the last 3 months before field tests realization.
  FEV1 will be assessed with non invasive spirometry.
Correlation between number of repetitions (STS Test) and number of exacerbations / year. | Number of exacerbations / year will assess the number of exacerbations in the last year before inclusion and will be assessed during the initial survey in the hour before field test realization.
Differences in dyspnea and muscular fatigue. | These outcomes will be assessed during both field tests. These tests will be separate by a 30 minutes rest period. Date will be collected at the end of each test up to 15 minutes.
  These outcomes will be assessed using Modified Borg Scale (0-10 points)
Differences in Heart Rate. | These outcomes will be assessed during both field tests. These tests will be separate by a 30 minutes rest period. Date will be collected at the end of each test up to 15 minutes.
  These outcomes will be assessed using pulse oximetry.
Differences in Respiratory Rate. | These outcomes will be assessed during both field tests. These tests will be separate by a 30 minutes rest period. Date will be collected at the end of each test up to 15 minutes
  These outcomes will be assessed using pulse oximetry.
Differences in Oxygen Saturation. | These outcomes will be assessed during both field tests. These tests will be separate by a 30 minutes rest period. Date will be collected at the end of each test up to 15 minutes.
  These outcomes will be assessed using pulse oximetry.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Le Roux, MD, Study Director — Groupe Hospitalier du Havre
Locations (3):
- France (3):
  - Hôpital Côte de Nacre, Caen
  - Le Havre Hospital, Le Havre
  - CHU de Rouen, Rouen

REFERENCES:
- [Background] Radtke T, Puhan MA, Hebestreit H, Kriemler S. The 1-min sit-to-stand test--A simple functional capacity test in cystic fibrosis? J Cyst Fibros. 2016 Mar;15(2):223-6. doi: 10.1016/j.jcf.2015.08.006. Epub 2015 Sep 9. PMID 26363563
- [Background] Ozalevli S, Ozden A, Itil O, Akkoclu A. Comparison of the Sit-to-Stand Test with 6 min walk test in patients with chronic obstructive pulmonary disease. Respir Med. 2007 Feb;101(2):286-93. doi: 10.1016/j.rmed.2006.05.007. Epub 2006 Jun 27. PMID 16806873
- [Background] Hussey J, Gormley J, Leen G, Greally P. Peripheral muscle strength in young males with cystic fibrosis. J Cyst Fibros. 2002 Sep;1(3):116-21. doi: 10.1016/s1569-1993(02)00074-7. PMID 15463817
- [Derived] Combret Y, Boujibar F, Gennari C, Medrinal C, Sicinski S, Bonnevie T, Gravier FE, Laurans M, Marguet C, Le Roux P, Lamia B, Prieur G, Reychler G. Measurement properties of the one-minute sit-to-stand test in children and adolescents with cystic fibrosis: A multicenter randomized cross-over trial. PLoS One. 2021 Feb 12;16(2):e0246781. doi: 10.1371/journal.pone.0246781. eCollection 2021. PMID 33577586